CLINICAL TRIAL: NCT05093803
Title: Study of Physical and Physiological Changes Through the Use of a Mobile App That Promotes Healthy Habits
Brief Title: Improvement of Physical and Physiological Parameters Through the Use of a Mobile App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Assistant Professor, University of Alicante
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: UA-2021-03-27
Record Dates: First submitted 2021-09-30; First posted 2021-10-26 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Hypertension; Diet, Healthy; Body Weight; Obesity; Cholesterol; Lipidosis; Machine Learning
MeSH Terms: conditions — Hypertension; Body Weight; Obesity; Lipidoses | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (Active Comparator): Recommendations on healthy eating habits based on the Mediterranean diet and moderate physical activity.
  Interventions: Behavioral: CONTROL GROUP
- APP GROUP (Experimental): Recommendations on healthy eating habits based on the Mediterranean diet and moderate physical activity through the use of an app based on machine learning, so they have constant stimuli for the improvement of the parameters.
  Interventions: Behavioral: HEALTH APP GROUP

INTERVENTIONS:
Behavioral: CONTROL GROUP — Intervention based on measurements of health parameters before and after providing participants with personalized dietary and physical activity recommendations.
  Arms: CONTROL GROUP
Behavioral: HEALTH APP GROUP — Use of a mobile application based on machine learning with the aim of improving health parameters and body composition.
  Specific diet program and moderate physical activity, all guided and mediated by a mobile application. As well as the recording and monitoring of periodic evaluations of health indicators.
  Other Names: Nutritional and physical activity intervention through the use of an app.
  Arms: APP GROUP

SUMMARY:
To investigate the health effects of a new mobile application (app) for prevention and personalized treatment in people with chronic cardiovascular pathologies associated with body composition.

DETAILED DESCRIPTION:
Scientific evidence has shown that the adoption of the Mediterranean diet is a protective factor against the appearance of several types of cancer, cardiovascular diseases, aging and obesity due to the amount of nutrients with anti-cancer, anti-inflammatory and anti-obesity properties that jointly contribute to the maintenance of health status. The antitumor effects of the Mediterranean diet are mainly due to the combination of antioxidant elements, fiber and polyunsaturated fats. Therefore, this dietary pattern is essential as a preventive measure against the onset of cancer and other chronic diseases, but also to reduce health care costs.

Monitoring physical activity should be considered as a central factor when addressing precision nutrition. Perform physical activity and exercise, as they are key components of energy expenditure and balance, in addition, structural changes occur in muscles, increase in the number of mitochondria in fiber, secretion of metabolically beneficial hormones with reversal of muscle insulin resistance and reduction of hepatic lipogenesis. Regardless of intensity, short-term exercise has been shown to improve adiposity and insulin sensitivity, which may help reduce metabolic risk. Boutcher et al. also demonstrated that intermittent aerobic and anaerobic exercise performed at an intensity >70% of maximal oxygen uptake significantly reduces ambulatory and office blood pressure in hypertensive individuals.

The development of this app aims, through self-management and visualizing the altered parameters and how they will evolve in your body in the short, medium and long term, to increase the population's commitment to these pathologies, in order to improve their health.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 21 years of age

Exclusion Criteria:

* Volunteers who do not have access to a smartphone.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
WEIGHT WEIGHT WEIGHT WEIGHT WEIGHT | 24 months
  The weight of the subjects will be obtained using the TANITA (Tokyo, Japan).
HEIGHT | 24 months
  The height of the subjects will be measured with the SECA 123 stadiometer (Hamburg, Germany).
WAIST CIRCUMFERENCE | 24 months
  The kinanthropometric evaluation is based on the methodology proposed for the restricted profile by the International Society for the Development of Kinanthropometry (ISAK). The material used to measure the perimeters will be a tape.
HIP CIRCUMFERENCE | 24 months
  The kinanthropometric evaluation is based on the methodology proposed for the restricted profile by the International Society for the Development of Kinanthropometry (ISAK). The material used to measure the perimeters will be a tape.
CHOLESTEROL | 24 months
  The blood cholesterol level is obtained through a blood test.
TRIGLICERIDES | 24 months
  The blood triglicerides level is obtained through a blood test.
BLOOD PREASURE | 24 months
  Measurement of blood pressure (systolic and diastolic) with a digital tensiometer.
FAT MASS | 24 months
  Assessment of body composition using the TANITA (Tokyo, Japan) validated bioimpedance scale to obtain the results of fat mass.
LEAN BODY MASS | 24 months
  Assessment of body composition using the TANITA (Tokyo, Japan) validated bioimpedance scale to obtain the results of lean body mass.
VISCERAL FAT | 24 months
  Assessment of body composition using the TANITA (Tokyo, Japan) validated bioimpedance scale to obtain the results of visceral fat.
HEART RATE | 24 months
  Heart rate measurement is performed with an activity wristband.
TROPONIN I | 24 months
  The troponin I level is obtained through a blood test.
BLOOD TROPONIN T LEVELS | 24 months
  The troponin I level is obtained through a blood test.
Broadband ultrasonic attenuation, BUA | 24 months
  The measurement of the ultrasonic band attenuation (BUA) by the traversed bone tissue (calcaneus) is performed using the GE Achilles Insight device.
Ultrasonic wave propagation speed, SOS | 24 months
  The measurement of ultrasonic wave propagation speed (SOS) by the traversed bone tissue (calcaneus) is performed using the GE Achilles Insight device.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Sánchez Sánchez, Full, Principal Investigator — European University of Madrid
Locations (1):
- Nutrición Selecta, Elche, Alicante, Spain